CLINICAL TRIAL: NCT04773509
Title: Effect of Intraoperative Paravertebral Block on Postoperative Pain and Recovery in Patients Undergoing Mechanical Correction for Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2020-1467
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2021-07

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Randomly selected patients of the PVB group are performed PVB with 0.2% ropivacaine on both sides. In contrast, PVB are not performed in the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, and outcomes assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVB group (Active Comparator): Patients of the PVB group are performed PVB with 0.2% ropivacaine on both sides
  Interventions: Procedure: Paravertebral block
- Control group (No Intervention): PVB are not performed in the control group.

INTERVENTIONS:
Procedure: Paravertebral block — Randomly selected patients of the PVB group are performed PVB with 0.2% ropivacaine on both sides.
  Arms: PVB group

SUMMARY:
Pain management after scoliosis surgery is challenging for the anesthesiologists. This surgery causes severe postoperative pain and patients undergoing these operations are children or adolescents who are increased pain sensation compared with adults. Therefore, we aim to evaluate whether intraoperative paravertebral block (PVB) decreases postoperative pain in these patients. Thirty-two patients scheduled for mechanical correction due to scoliosis will be divided into PVB (n=16) and control (n=16) groups. Randomly selected patients of the PVB group are performed PVB with 0.2% ropivacaine on both sides. In contrast, PVB are not performed in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mechanical correction

Exclusion Criteria:

* The subjects who cannot communicate
* The subject is a foreigner or illiterate

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Pain score | 6 hours after the end of surgery
  visual analog scale (VAS) (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lee, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No